CLINICAL TRIAL: NCT02948426
Title: Phase 1 Study of Intraperitoneal Infusion of Autologous Monocytes With Sylatron (Peginterferon Alfa-2b) and Actimmune (Interferon Gamma-1b) in Women With Recurrent or Refractory Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer
Brief Title: Intraperitoneal Infusion of Autologous Monocytes With Sylatron (Peginterferon Alfa-2b) and Actimmune (Interferon Gamma-1b) in Women With Recurrent or Refractory Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was closed to accrual due to lack of drug supply.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stanley Lipkowitz, MD, PhD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170011; 17-C-0011
Record Dates: First submitted 2016-10-27; First posted 2016-10-28 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cancer
Keywords: Immunotherapy; Adoptive Cell Therapy; Carcinomatosis; CA125
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma | interventions — interferon gamma-1b; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) (Experimental): Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml). The autologous monocytes cell product in 250ml total volume of investigational combination (monocytes + ACTIMMUNE + SYLATRON) is infused via the intraperitoneal catheter over 30-60 min +/- 10 min every 28 days +/- 7 days until disease progression, limiting toxicity, intercurrent medical issues, or patient withdrawal.
  Interventions: Biological: Autologous Monocytes + ACTIMMUNE + SYLATRON
- Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) (Experimental): Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml). The autologous monocytes cell product in 250ml total volume of investigational combination (monocytes + ACTIMMUNE + SYLATRON) is infused via the intraperitoneal catheter over 30-60 min +/- 10 min every 28 days +/- 7 days until disease progression, limiting toxicity, intercurrent medical issues, or patient withdrawal.
  Interventions: Biological: Autologous Monocytes + ACTIMMUNE + SYLATRON
- Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) (Experimental): Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml). The autologous monocytes cell product in 250ml total volume of investigational combination (monocytes + ACTIMMUNE + SYLATRON) is infused via the intraperitoneal catheter over 30-60 min +/- 10 min every 28 days +/- 7 days until disease progression, limiting toxicity, intercurrent medical issues, or patient withdrawal.
  Interventions: Biological: Autologous Monocytes + ACTIMMUNE + SYLATRON
- Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml) (Experimental): Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml). The autologous monocytes cell product in 250ml total volume of investigational combination (monocytes + ACTIMMUNE + SYLATRON) is infused via the intraperitoneal catheter over 30-60 min +/- 10 min every 28 days +/- 7 days until disease progression, limiting toxicity, intercurrent medical issues, or patient withdrawal.
  Interventions: Biological: Autologous Monocytes + ACTIMMUNE + SYLATRON
- EX1 Dose Expansion Arm (Experimental): 10 additional patients will be treated at the maximum tolerated dose (MTD)
  Interventions: Biological: Autologous Monocytes + ACTIMMUNE + SYLATRON

INTERVENTIONS:
Biological: Autologous Monocytes + ACTIMMUNE + SYLATRON — The autologous monocytes cell product in 250ml total volume of investigational combination (monocytes + ACTIMMUNE + SYLATRON) is infused via the intraperitoneal catheter over 30-60 min +/- 10 min every 28 days +/- 7 days until disease progression, limiting toxicity, intercurrent medical issues, or patient withdrawal. Dosing is based on a dose escalation design including an expansion cohort at the maximum tolerated dose (MTD).

SUMMARY:
Ovarian cancer is a leading cause of cancer death in women. Monocytes are white blood cells that slow tumor growth. Interferons (IFNs) are molecules that help immune cells fight cancer. Researchers want to stimulate monocytes with IFNs. They want to test if these stimulated monocytes combined with the drugs Sylatron and Actimmune can shrink tumors and slow the progression of cancer.

Objective:

To test how well IFN stimulated monocytes, with Sylatron and Actimmune, kill tumor cells.

Eligibility:

Women ages 18 and older with certain ovarian, fallopian tube, or peritoneal cancers

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Scan

Results or sample from previous biopsy

Participants may have a tumor sample taken.

Participants who do not have a port will have a catheter placed inside the abdominal cavity. It will be used to give the treatment.

Participants will have visits for 4 days of each 28-day cycle. This includes overnight observation.

Participants with ascites fluid in their abdominal cavity will have it sampled twice.

Each cycle, participants will have:

Blood tests

Leukapheresis. Some blood is removed and put through a machine that separates out the monocytes. The rest of the blood is returned to the body.

Infusion of the monocytes and study drugs

Participants will have weekly phone calls in Cycle 1 and scans every 2 cycles.

Participants will continue treatment until they can no longer tolerate it or their cancer gets worse.

Participants will have a visit about 1 month after stopping treatment, then monthly phone calls.

DETAILED DESCRIPTION:
Background:

* Monocytes can differentiate into classic M1 (classically activated) macrophages inhibiting tumor proliferation and promoting natural killer (NK) cell differentiation.
* Human alpha interferons (interferon alfa, IFN-alpha), interferon gamma (IFN-gamma) and monocytes have strong anti-neoplastic response in vitro and in vivo
* IFN-alpha and IFN-gamma have been shown in early phase clinical trials to be safely administered intraperitoneally.
* Intraperitoneal monocytes alone or activated with IFN-gamma are safe and feasible as demonstrated in phase I clinical studies.
* We have shown that the combination of human monocytes, IFN-alpha2a and IFN-gamma1b, or pegylated IFN-alpha, act synergistically against tumor cells in vitro and in mouse models.

Objectives:

-To identify a maximum tolerated dose of intraperitoneal autologous monocytes and Sylatron(R) (Peginterferon alfa-2b) and Actimmune(R) (Interferon gamma-1b).

Eligibility:

* Advanced metastatic or unresectable epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer that is relapsed and resistant or refractory to prior platinum-based standard care systemic regimen.
* Patients must be off prior chemotherapy, radiation therapy, hormonal therapy or biological therapy for at least 4 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 and adequate organ and marrow function.

Design:

* This is an open label single arm phase I trial to determine the maximum tolerated dose of intraperitoneal monocytes and Sylatron(R) (Peginterferon alfa-2b) and Actimmune(R) (Interferon gamma-1b).
* Autologous monocytes obtained through apheresis will be mixed with Sylatron(R) (Peginterferon alfa-2b) and Actimmune(R) (Interferon gamma-1b) in a 3 + 3 dose escalation and administered intraperitoneally once every 28 days. A new product will be manufactured for each treatment cycle.
* Once the maximum tolerated dose is obtained, an expansion cohort will be enrolled to better quantify response rate and time to disease progression.
* Research samples including peripheral blood and ascites will be obtained prior to the initiation of study therapy andprior to the start of each cycle. Tissue biopsies will be obtained in the dose expansion phase to characterize the immune infiltration.
* Patients will be evaluated every 2 cycles for response using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and every cycle for safety using Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed advanced metastatic or unresectable epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer that is relapsed and resistant (recurred less than 6 months after chemotherapy) or refractory (progressed on chemotherapy) to prior platinum- and taxane-based standard care systemic regimen. Or patients who are eligible for aditional platinum therapy. Histopathologic diagnosis must be confirmed in the Laboratory of Pathology (LP), National Cancer Institute (NCI).
* Patients must have measurable or evaluable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* Patients must be at least 4 weeks from previous therapy (chemotherapy, hormonal therapy, and radiation therapy, immunotherapy and monoclonal antibodies, alternative therapy or investigational therapeutic agents). There is no limitation on the amount of prior therapies allowed. Patients with ovarian cancer 4 weeks from previous therapy have been found to have normal monocyte function (unpublished).
* Patients who have had cranial radiation therapy need to have completed it greater than or equal to 8 weeks prior to enrollment.
* Patients are permitted to receive investigational imaging agents while on study.
* Patients who have had major surgery must be fully recovered and require a recovery period of greater than or equal to 4 weeks prior to enrolling on study.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of intraperitoneal monocytes, interferon (IFN)-alpha 2 or IFN-gamma in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 70%).
* Adequate renal function, defined as serum creatinine less than or equal to 1.5 X upper limit of normal (ULN), or measured creatinine clearance greater than or equal to 60 mL/min/1.73m^2.
* Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilbert's syndrome, where bilirubin less than or equal to 5 mg/dl will be permitted. Gilbert's syndrome will be defined as elevated unconjugated bilirubin, with conjugated (direct) bilirubin within the normal range and less than 20% of the total. Total bilirubin will be permitted up to 5 mg/dl, if patients have historical readings consistent with the definition of Gilbert's syndrome prior to entering study.
* Adequate bone marrow function, defined as absolute neutrophil (ANC) greater than or equal to 1,500/mm^3 (greater than or equal to 1.5 X106/L), platelet count greater than or equal to 75,000/mm^3 (greater than or equal to 75 X10^6/L), and hemoglobin greater than or equal to 8 g/dL (transfusion to obtain hemoglobin greater than or equal to 8 g/dL is allowed).
* The effects of intraperitoneal monocytes, IFN-alpha 2, and IFN-gamma on the developing human fetus are unknown. For this reason and because interferons based on animal data may cause fetal harm, women of child-bearing potential (excludes women with recurrent ovarian cancer) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents (with exception of imaging agents as indicated above in the inclusion criteria).
* Patients cannot have previously been treated with interferons (e.g., for chronic active hepatitis).
* Lack of recovery of prior adverse events to Grade less than or equal to 1 severity (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v 4.03) (except alopecia) due to therapy administered prior to the initiation of study drug dosing. Stable persistent grade 2 peripheral neuropathy may be allowed as determined on a case-bycase basis at the discretion of the Investigator as interferon has not been shown to cause or exacerbate peripheral neuropathy.
* Patients with active infection will not be eligible, but may become eligible once infection has resolved and at least 7 days have elapsed after antibiotics use was completed.
* Concomitant chronic (daily or almost daily for greater than or equal to 1 month prior) use of steroids or non-steroidal anti-steroidal anti-inflammatory drugs (NSAIDS).
* Patients with a recent history (within last 5 years) of autoimmune disease or inflammatory diseases will be excluded, because interferons may worsen these conditions. Exceptions will be allowed for vitiligo and hypothyroidism that has been stable on thyroid replacement medications for >6 weeks.
* Impaired cardiac function or clinically significant cardiac disease including the following:

  * New York Heart Association class III or IV congestive heart failure
  * Myocardial infarction within the last 12 months
  * Subjects known to have impaired left ventricular ejection fraction (LVEF) according to institutional standards
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to interferons or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations within the last 12 months that would limit compliance with study requirements. Patients with history of neuropsychiatric disorders or Major Depressive Disorder (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) definition: http://dsm.psychiatryonline.org/doi/full/10.1176/appi.books.9780890425596.dsm04) requiring medical treatment will not be eligible to enroll, based on the black box warning (SYLATRON (peginterferon alfa-2b) for injection, for subcutaneous use. Merck Sharp & Dohme Corp., a subsidiary of Merck & Co., Inc., Whitehouse Station, NJ). Exception to this is if patients experienced transient post-partum depression that resolved and patient has been off treatment for >10 years. Patients who are taking oral anti-depressants for normal sadness, bereavement, or grief will not be excluded.
* Pregnant women are excluded from this study because interferons based on animal data may cause fetal harm. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with interferons, breastfeeding should be discontinued if the mother is treated with intraperitoneal interferons. These potential risks may also apply to other agents used in this study.
* Patients on combination antiretroviral therapy for the treatment of HIV are ineligible because of the potential for pharmacokinetic interactions with interferons alfa and gamma.
* Patients receiving any medications or substances that are potent inhibitors or inducers of Cytochrome P450 1A2 (CYP1A2) or Cytochrome P450 2D6 (CYP2D6) are ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Lipkowitz, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Johnson CL, Green DS, Zoon KC. Human monocytes in the presence of interferons alpha2a and gamma are potent killers of serous ovarian cancer cell lines in combination with paclitaxel and carboplatin. J Interferon Cytokine Res. 2015 Jan;35(1):55-62. doi: 10.1089/jir.2014.0057. Epub 2014 Jul 28. PMID 25068849
- [Background] Soderquest K, Powell N, Luci C, van Rooijen N, Hidalgo A, Geissmann F, Walzer T, Lord GM, Martin-Fontecha A. Monocytes control natural killer cell differentiation to effector phenotypes. Blood. 2011 Apr 28;117(17):4511-8. doi: 10.1182/blood-2010-10-312264. Epub 2011 Mar 9. Erratum In: Blood. 2013 Sep 26;122(13):2290. PMID 21389319
- [Background] Artis D, Spits H. The biology of innate lymphoid cells. Nature. 2015 Jan 15;517(7534):293-301. doi: 10.1038/nature14189. PMID 25592534
- [Background] Phase 1 study of intraperitoneal infusion of autologous monocytes with peginterferon alfa-2b and interferon gamma-1b in women with recurrent or refractory ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. By: Nunes, Ana Tablante; Green, Daniel; Ekwede, Irene; et al. Conference: 53rd Annual Meeting of the American-Society-of-Clinical-Oncology (ASCO) Location: Chicago, IL Date: JUN 02-06, 2017 Sponsor(s): Amer Soc Clin Oncol JOURNAL OF CLINICAL ONCOLOGY Volume: 35 Supplement: 15 Meeting Abstract: TPS3092 Published: MAY 20 2017
- [Background] Production of autologous monocytes stimulated ex vivo with peg-interferon alfa 2b and interferon gamma 1b for intraperitoneal administration in phase I clinical trial. By: Duemler, Anna; Green, Daniel S.; Highfill, Steven L.; et al. Conference: ASCO-SITC Clinical Immuno-Oncology Symposium Location: San Francisco, CA Date: FEB 28-MAR 02, 2019 Sponsor(s): ASCO; SITC JOURNAL OF CLINICAL ONCOLOGY Volume: 37 Issue: 8 Supplement: S Meeting Abstract: 5 Published: MAR 10 2019
- [Background] Green DS, Nunes AT, David-Ocampo V, Ekwede IB, Houston ND, Highfill SL, Khuu H, Stroncek DF, Steinberg SM, Zoon KC, Annunziata CM. A Phase 1 trial of autologous monocytes stimulated ex vivo with Sylatron(R) (Peginterferon alfa-2b) and Actimmune(R) (Interferon gamma-1b) for intra-peritoneal administration in recurrent ovarian cancer. J Transl Med. 2018 Jul 16;16(1):196. doi: 10.1186/s12967-018-1569-5. PMID 30012146
- [Background] Green DS, Nunes AT, Tosh KW, David-Ocampo V, Fellowes VS, Ren J, Jin J, Frodigh SE, Pham C, Procter J, Tran C, Ekwede I, Khuu H, Stroncek DF, Highfill SL, Zoon KC, Annunziata CM. Production of a cellular product consisting of monocytes stimulated with Sylatron(R) (Peginterferon alfa-2b) and Actimmune(R) (Interferon gamma-1b) for human use. J Transl Med. 2019 Mar 14;17(1):82. doi: 10.1186/s12967-019-1822-6. PMID 30871636
- [Result] First-in-human phase I study of intraperitoneally administered interferon-activated autologous monocytes in platinum-resistant or refractory ovarian cancer By: Cole, Christopher Browning; Annunziata, Christina M. Conference: ASCO-SITC Clinical Immuno-Oncology Symposium Location: Orlando, FL Date: FEB 06-08, 2020 Sponsor(s): Amer Soc Clin Oncol; Soc Immunotherapy Canc JOURNAL OF CLINICAL ONCOLOGY Volume: 38 Issue: 5 Supplement: S Meeting Abstract: 1 Published: FEB 10 2020
- [Derived] Kamat K, Krishnan V, Berek JS, Dorigo O. Cell-based immunotherapy in gynecologic malignancies. Curr Opin Obstet Gynecol. 2021 Feb 1;33(1):13-18. doi: 10.1097/GCO.0000000000000676. PMID 33278077
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0011.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled on the EX 1 Dose Expansion Arm/Group.
Period: Overall Study
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml)
Started | 3 | 6 | 3 | 6
Completed | 3 | 6 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml) | Total
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 1 | 4 | 12
  >=65 years | 1 | 1 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.77 (9.16) | 58.17 (8.84) | 62.33 (9.22) | 60.67 (12.47) | 60.63 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 6 | 18
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 3 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3
  White | 1 | 5 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 3 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Maximum Tolerated Dose of Intraperitoneal Autologous Monocytes
Description: Maximum Tolerated Dose of intraperitoneal autologous monocytes.
Time Frame: Cycle 1 Day 28
Measure: Number; unit: Cells
Groups:
- All Participants On Dose Level 1 Through Dose Level 4: Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Dose Level 2 - Sylatron 25µg (0.1µg/ml); Dose Level 3 - Sylatron 25mcg; Dose Level 4 - Sylatron 250mcg
Arm/Group | All Participants On Dose Level 1 Through Dose Level 4
Number analyzed (Participants) | 18
Cells | 750000000

2. Primary Outcome: Overall Maximum Tolerated Dose of Sylatron (Peginterferon Alpha-2b)
Description: Maximum Tolerated Dose of Sylatron (Peginterferon alpha-2b).
Time Frame: Cycle 1 Day 28
Measure: Number; unit: mcg
Arm/Group | All Participants On Dose Level 1 Through Dose Level 4
Number analyzed (Participants) | 18
mcg | 250

3. Primary Outcome: Overall Maximum Tolerated Dose of Actimmune (Interferon Gamma-1b)
Description: Maximum Tolerated Dose of Actimmune (Interferon gamma-1b).
Time Frame: Cycle 1 Day 28
Measure: Number; unit: mcg
Groups:
- All Participants On Dose Level 1 Through Dose Level 4: Dose Level 1 - Actimmune 5mcg (0.02µg/ml); Dose Level 2 - Actimmune 5mcg (0.02µg/ml); Dose Level 3 - Actimmune 5mcg; Dose Level 4 - Actimmune 50mcg
Arm/Group | All Participants On Dose Level 1 Through Dose Level 4
Number analyzed (Participants) | 18
mcg | 50

4. Secondary Outcome: Number of Participants With a Response
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Participants were evaluated for response by radiographic imaging every 8 weeks, up to 80 weeks
Population: One participant is not included in the analysis because the participant was not evaluable for response in dose level 1. The participant came off study due to inability to replace her IP catheter (became ineligible) after cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml)
Number analyzed (Participants) | 2 | 6 | 3 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 1
  Stable Disease | 0 | 2 | 1 | 2
  Progressive Disease | 1 | 4 | 2 | 3

5. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to progression, censored at date last known progression-free for those who have not progressed. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study
Time Frame: Participants were assessed every 4 weeks by physical exam and 8 weeks by radiographic imaging for disease progression, up to 10 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml)
Number analyzed (Participants) | 3 | 6 | 3 | 6
Months | 3.7 [1 to 8] | 3.2 [1 to 10] | 2.0 [1 to 3] | 3.7 [1 to 10]

6. Other Pre Specified Outcome: Number of Participants With Serious or Non-serious (Any) Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 10 months and 11 days for dose level 1,12 months and 1 day for dose level 2, 11 months and 4 days for dose level 3, and 12 months and 6 days for dose level 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml)
Number analyzed (Participants) | 3 | 6 | 3 | 6
Participants | 3 | 6 | 3 | 6

7. Other Pre Specified Outcome: Number of Participants With a Grade 3 or Higher Dose-Limiting Toxicity (DLT)
Description: DLT is defined as an laboratory abnormality or adverse drug reaction (ADR) according to the Common Terminology Criteria for Adverse Events (CTCAE), such as any grade 4 immune mediated adverse event attributed to local tumor response, any grade ≥3 colitis, grade 3 or 4 noninfectious pneumonitis, and any > grade 2 cardiac toxicity which dose not resolve to grade 1 within 3 days of initiation of maximum supportive care that is possibly, probably, or definitely related to the combination of drug. Grade 3 adverse event is severe or medically significant but not immediately life-threatening, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: Cycle 1 Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml)
Number analyzed (Participants) | 3 | 6 | 3 | 6
Participants | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 10 months and 11 days for dose level 1,12 months and 1 day for dose level 2, 11 months and 4 days for dose level 3, and 12 months and 6 days for dose level 4.
Arm/Group | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml)
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/6 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 6/6 | 2/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) (N=3) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) (N=6) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) (N=3) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml) (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Sylatron 25µg (0.1 µg/ml); Actimmune 5mg (0.02µg/ml) (N=3) | Dose Level 2 - Monocytes (75x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) (N=6) | Dose Level 3 - Monocytes (750x10^6); Sylatron 25µg (0.1µg/ml); Actimmune 5mg (0.02µg/ml) (N=3) | Dose Level 4 - Monocytes (750x10^6); Sylatron 250µg (1µg/ml); Actimmune 50mg (0.2µg/ml) (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 3 (6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 3 (3) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 4 (7) | 2 (4) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (15) | 6 (25) | 2 (10) | 5 (19)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 2 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, SEM III/VI (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (5) | 4 (9) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (6)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (4)
Flashing lights (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, 3Lightheaded (after hydromorphone) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Decrease performance status (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Lightheadedness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Night sweats (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5) | 6 (19) | 1 (1) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (12) | 1 (1) | 2 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (10) | 5 (14) | 2 (4) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (6) | 3 (8) | 1 (2) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 2 (6) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (7) | 6 (28) | 3 (9) | 6 (28)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (2) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 2 (3) | 2 (5) | 1 (3) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders - Other, arterial bleeding (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (6)
White blood cell decreased (Investigations) | 1 (2) | 1 (4) | 0 (0) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT02948426/Prot_SAP_003.pdf
  • Informed Consent Form (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT02948426/ICF_004.pdf